CLINICAL TRIAL: NCT03629171
Title: Phase II Study of CPX-351 in Combination With Venetoclax in Patients With Acute Myeloid Leukemia (AML)
Brief Title: Liposome-encapsulated Daunorubicin-Cytarabine and Venetoclax in Treating Participants With Relapsed, Refractory or Untreated Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-1055; NCI-2018-01589 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-1055 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-08-09; First posted 2018-08-14 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — CPX-351; Injections; Daunorubicin; Cytarabine; Liposomes; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (CPX-351, venetoclax) (Experimental): INDUCTION: Participants receive liposome-encapsulated daunorubicin-cytarabine IV over 90 minutes on days 1, 3, and 5 of cycle 1 and on days 1 and 3 of cycle 2. Participants also receive venetoclax PO QD on days 2-21. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION: Participants receive liposome-encapsulated daunorubicin-cytarabine IV over 90 minutes on days 1 and 3 and venetoclax PO QD on days 2-21. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Liposome-encapsulated Daunorubicin-Cytarabine; Drug: Venetoclax

INTERVENTIONS:
Drug: Liposome-encapsulated Daunorubicin-Cytarabine — Given IV
  Other Names: CPX-351; Cytarabine-Daunorubicin Liposome for Injection; Daunorubicin and Cytarabine (Liposomal); Liposomal AraC-Daunorubicin CPX-351; Liposomal Cytarabine-Daunorubicin; Liposome-encapsulated Combination of Daunorubicin and Cytarabine; Vyxeos
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase II trial studies how well liposome-encapsulated daunorubicin-cytarabine and venetoclax work in treating participants with acute myeloid leukemia that has come back (relapsed), does not respond to treatment (refractory), or has not been treated (untreated). Drugs used in chemotherapy, such as liposome-encapsulated daunorubicin-cytarabine and venetoclax, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the efficacy (complete remission [CR], complete remission without blood count recovery [CRi], complete remission without platelet recovery [CRp]) of liposome-encapsulated daunorubicin-cytarabine (CPX-351) in combination with venetoclax in patients with acute myeloid leukemia (AML).

SECONDARY OBJECTIVES:

I. To assess safety of CPX-351 in combination with venetoclax in patients with AML.

II. To assess the event free survival (EFS) and overall survival (OS) in patients with AML.

EXPLORATORY OBJECTIVE:

I. To explore biomarkers of response and resistance in AML treated with CPX-351 and venetoclax.

OUTLINE: This is a dose-escalation study of venetoclax.

INDUCTION: Participants receive liposome-encapsulated daunorubicin-cytarabine intravenously (IV) over 90 minutes on days 1, 3, and 5 of cycle 1 and on days 1 and 3 of cycle 2. Participants also receive venetoclax orally (PO) once daily (QD) on days 2-21. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION: Participants receive liposome-encapsulated daunorubicin-cytarabine IV over 90 minutes on days 1 and 3 and venetoclax PO QD on days 2-21. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up at 30 days and then every 3 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* For the lead in phase: Patients >= 18 years of age with a diagnosis of relapsed and/or refractory AML will be eligible. Patients who have had prior treatment with venetoclax will be allowed to participate in the lead in phase and cohort A
* For the dose expansion cohort A (relapsed/refractory [R/R] AML): Patients >= 18 years of age with a diagnosis of relapsed and/or refractory AML will be eligible
* For the dose expansion cohort B (de novo AML): Patients >= 18 years to 69 years of age; patients in this cohort must have received no prior therapy for AML
* Prior therapy with hydroxyurea, hematopoietic growth factors, or tretinoin (ATRA) (for emergency use for stabilization) is allowed with no washout. A cumulative dose of ara-C of up to 3 g for emergency stabilization in patients with rapidly proliferating disease is also allowed provided it was administered > 48 hrs prior to enrollment
* Bilirubin =< 2 mg/dL
* Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) =< 3 x upper limit of normal (ULN) or < 5 x ULN if related to leukemic involvement
* Creatinine =< 1.5 x ULN
* Known cardiac ejection fraction of > or = 45% within the past 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* A negative urine or serum pregnancy test is required within 1 week for all women of childbearing potential prior to enrolling on this trial. A woman of childbearing potential is defined as a woman who has not been naturally postmenopausal for at least 12 consecutive months, or who had no previous surgical sterilization
* Patient must have the ability to understand the requirements of the study and signed informed consent. A signed informed consent by the patient or his legally authorized representative is required prior to their enrollment on the protocol

Exclusion Criteria:

* Pregnant women are excluded from this study because the agents used in this study have the potential for teratogenic or abortifacient effects. Because there is a potential risk for adverse events in nursing infants secondary to treatment of the mother with the chemotherapy agents, breastfeeding should also be avoided
* Uncontrolled intercurrent illness including, but not limited to active uncontrolled infection, symptomatic congestive heart failure (New York Heart Association [NYHA] class III or IV), unstable angina pectoris, clinically significant cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patient with documented hypersensitivity to any of the components of the chemotherapy program
* Patients with acute promyelocytic leukemia (M3) or core-binding factor AML
* Patients with active central nervous system (CNS) leukemia are excluded since the antileukemia activity of the treatment components against CNS leukemia are not known
* Men and women of childbearing potential who do not practice contraception. Women of childbearing potential and men must agree to use contraception prior to study entry and for the duration of study participation
* Prior treatment with CPX-351 or venetoclax. Patients with prior treatment with venetoclax will be allowed in patients with relapsed/refractory (R/R) disease including those in the lead-in phase as well as those in cohort A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2018-10-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Achievement of composite complete remission | Up to 3 cycles (84 days)
  Defined as complete remission/complete remission without blood count recovery/complete remission without platelet recovery. Will be monitored simultaneously using the Bayesian approach of Thall, Simon, Estey. Will be estimated along with the 95% credible interval.
Incidence of adverse events | Up to 28 days
  Will be monitored simultaneously using the Bayesian approach of Thall, Simon, Estey. Will be summarized using descriptive statistics such as mean, standard deviation, median and range. Safety data will be summarized by category, severity and frequency.

SECONDARY OUTCOMES:
Event-free survival | Number of days from the date of treatment initiation up to 1 year
  Will be estimated using the method of Kaplan and Meier. Comparisons of time-to-event endpoints by important subgroups will be made using the log-rank tests.
Overall survival | Time from treatment start till death or last follow-up, assessed up to 1 year
  Will be estimated using the method of Kaplan and Meier. Comparisons of time-to-event endpoints by important subgroups will be made using the log-rank tests.
Biomarker changes | Baseline up to 1 year
  The comparison regarding biomarkers between response and non-response will be conducted by two-sample t-test if the data is normally distributed, otherwise Wilcoxon rank sum test will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Tapan M Kadia, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Kadia TM, Jen WY, Bataller A, Bazinet A, Borthakur G, Jabbour E, Qiao W, Short NJ, Takahashi K, Issa GC, DiNardo CD, Montalban-Bravo G, Pemmaraju N, Tran A, Bharathi V, Loghavi S, Alousi AM, Popat U, Daver NG, Ravandi F, Kantarjian HM. A Phase 2 Trial of CPX-351 Combined With Venetoclax in Relapsed or Refractory Acute Myeloid Leukemia. Am J Hematol. 2025 Aug;100(8):1365-1373. doi: 10.1002/ajh.27723. Epub 2025 May 22. PMID 40401707
- See also: MD Anderson Cancer Center — http://www.mdanderson.org